CLINICAL TRIAL: NCT07301411
Title: An Exploratory Clinical Trial Evaluating Navigational Bronchoscopy System and Bronchoscope and Accessories in Combination With Cryoablation Therapy Device for the Treatment of Lung Malignancies
Brief Title: Exploratory Trial of Navigational Bronchoscopy-Guided Cryoablation in Lung Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Puli Ark Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-002
Record Dates: First submitted 2025-12-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Malignancies
Keywords: Navigational Bronchoscopy System; Lung Malignancies; Cryoablation
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- An exploratory clinical trial with two cohorts (Experimental): Cohort1: Enrolled subjects will undergo bronchoscopy-guided cryoablation procedure for treating malignant lung nodules in Shanghai Chest Hospital, China.
  Cohort2: Enrolled subjects will undergo bronchoscopy-guided cryoablation procedure for treating malignant lung nodules at the Prince of Wales Hospital of the Chinese University of Hong Kong.
  The two cohorts differ in the manufacturer of the bronchoscope and accessories used at each site.
  Interventions: Device: Cryoablation Therapy

INTERVENTIONS:
Device: Cryoablation Therapy — Navigational Bronchoscopy System and Bronchoscope and Accessories in Combination with Cryoablation Therapy Device.
  Other Names: Navigational Bronchoscopy System; Bronchoscope and Accessories; Cryoablation Therapy Device

SUMMARY:
This clinical trial is an exploratory clinical trial with two cohorts:

Cohort 1: aiming to conduct a preliminary evaluation of the effectiveness and safety of the Navigational Bronchoscopy System and the Bronchoscope and Accessories (manufactured by Noah) in combination with the cryoablation therapy devices for the treatment of lung malignancies.

Cohort 2: aiming to conduct a preliminary evaluation of the effectiveness and safety of the Navigational Bronchoscopy System and the Bronchoscope and Accessories (manufactured by Puli Ark) in combination with the cryoablation therapy devices for the treatment of lung malignancies.

The overall objective of this study is to conduct a preliminary evaluation of the effectiveness and safety of navigational bronchoscopy - guided cryoablation therapy of the lungs through the above two cohorts.

DETAILED DESCRIPTION:
This clinical trial adopts a prospective, dual-center, exploratory design, aiming for a preliminary evaluation of the effectiveness and safety of the investigational medical devices Navigational Bronchoscopy System and Bronchoscope and Accessories in combination with cryoablation therapy device for the treatment of lung malignancies. The clinical trial is planned to be conducted at two clinical trial institutions, with approximately 40 subjects enrolled in total. Subjects who have signed the informed consent form (ICF), meet the conditions for this trial, meet all inclusion criteria and do not meet any exclusion criteria will be included in this study. Enrolled subjects will receive the investigational medical devices Navigational Bronchoscopy System and Bronchoscope and Accessories in combination with cryoablation therapy device for the treatment of lung malignancies on Day 0. Subjects will undergo safety and effectiveness evaluations on the following timelines: Day 1 post-treatment (within 24 hours after treatment), 1 month post-treatment (Day 30 ± 7 days after treatment), and 3 months post-treatment (Day 90 ± 14 days after treatment). After completing the follow-up visit at 3 months post-treatment (Day 90 ± 14 days post-treatment), investigators at each study site, at their discretion, will conduct subsequent treatments based on routine medical practice, and will continue follow-up to 12 months post-treatment and record relevant clinical data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old (inclusive), male or female;
2. Primary peripheral lung cancer, with pre-treatment staging examination indicating clinical stage T1N0M0, IA (including new onset and multiple primary lesions after treatment); or metastatic lung tumor, with the primary lesion completely removed or well controlled;
3. The maximum diameter of the tumor is ≤3 cm;
4. The number of tumors is ≤3 (no limit for multiple primary lung cancer subjects);
5. Subjects who decline or are deemed unsuitable for surgery per multidisciplinary team's discretion;
6. Subjects who decline or are deemed unsuitable for radiotherapy per investigator's discretion;
7. Subjects whose lesions to be ablated are assessed to be feasible for bronchoscopy-guided cryoablation per investigator's discretion;
8. Subjects who are willing to participate in the study and sign the written informed consent.

Exclusion Criteria:

1. Subjects with diffuse lesions in both lungs whose condition cannot be improved by ablation treatment;
2. Subjects whose examination within 1 month prior to treatment suggests intrathoracic lymph node metastasis or extrapulmonary metastasis (except for those whose extrapulmonary metastasis is controlled by local treatment);
3. With reference to the Guidelines for the Application of Diagnostic Flexible Bronchoscopy for Adults (2019 Edition) [1], subjects with contraindications for bronchoscopy, such as acute myocardial infarction (within 4 weeks), active massive hemoptysis, platelet count < 60×109/L, malignant arrhythmia, unstable angina, severe cardiopulmonary insufficiency, hypertensive crisis, severe pulmonary hypertension, intracranial hypertension, acute cerebrovascular events (i.e. cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, intracranial venous thrombosis, etc.), aortic dissection, aortic aneurysm, and systemic extreme failure;
4. Subjects who are using antiplatelet or anticoagulant drugs and cannot be properly managed before treatment (properly managed including clopidogrel terminated 7 days before treatment, ticagrelor terminated 5 days before treatment, warfarin terminated 5 days before treatment, low molecular weight heparin terminated 24 hours before treatment, etc.);
5. Subjects with severe bleeding tendency, uncorrectable coagulation dysfunction;
6. Subjects with electrically or magnetically activated devices implanted or metallic implants (non-titanium);
7. Subjects with other tumors and extensive metastasis, with an expected survival of less than 12 months;
8. Poor general condition (e.g. systemic multiple metastases, severe infection, high fever), infectious and radioactive inflammation around the focus, obvious cachexia, serious dysfunction of important organs, severe anemia and nutritional metabolism disorder that cannot be improved in a short time;
9. The subjects with Eastern Cooperative Oncology Group (ECOG) performance status score of >2 (See Appendix 1 for details of ECOG scoring criteria);
10. Subjects having received radiotherapy within the past 6 months for the lesion to be ablated;
11. Subjects expected to participate in any other experimental or invasive clinical study within 12 months of the ablation procedure;
12. Subjects with a history of active hepatitis B, active hepatitis C, human immunodeficiency virus (HIV) infection (known HIV1/2 antibody positive) or, in the investigator's judgment, conditions that may affect the subject's treatment;
13. Those with epilepsy, psychiatric history or cognitive impairment;
14. Pregnant, lactating women, and subjects who are unwilling to use reasonable contraception during the clinical trial;
15. Subjects who had participated or are participating in a drug clinical trial within 3 months (participants in non-interventional trials can be included), or who had participated or are participating in another medical device clinical trial within 1 month (participants in non-interventional trials can be included);
16. Other circumstances which are considered by the investigator not suitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate (ablation lesion level) | Immediately following the procedure (no more than 30 minutes after completion of all ablation deliveries)
  Definition of technical success: Immediately following the procedure (no more than 30 minutes after completion of all ablation deliveries), the cone-beam computerized tomography (CBCT) imaging (evaluated by treating investigator) shows that the target lesion is covered completely by the ablation zone (i.e., the ablation zone completely overlaps or encompasses target tumor plus an ablative margin (a minimum of 5 mm ablative margin).

SECONDARY OUTCOMES:
Technique efficacy rate at 3 months after treatment (ablation lesion level) | 3 months after ablation treatment
  Definition of technique efficacy rate: 3 months after ablation treatment, the percentage of target tumors successfully eradicated in the total number of lesions receiving ablation treatment.
Disease control rate | At 3 months follow-ups.
  Disease control rate is defined as the proportion of target ablated lesions that achieve complete ablation and incomplete ablation as assessed by imaging in the total number of ablated lesions at 3 months follow-ups.
Navigation success rate | During the cryoablation procedure
  Criteria for successful navigation: Navigation is considered successful if lesion arrival is confirmed by the navigation system and the distance between the bronchoscope and the margin of preoperative planning target is less than 2 cm, or the actual distance is judged by the investigator to be sufficient to complete the ablation and the ablation is successful. Otherwise, navigation is considered a failure.
Quality of life score | At screening period/baseline, 1 month post-treatment, and 3 months post-treatment follow-up
  Quality of life is scored by the European Organization for Research and Treatment of Cancer (EORCT) Quality of Life Questionnaire-Core 30 scale (QLQ-C30) at screening period/baseline, 1 month post-treatment, and 3 months post-treatment follow-up.
  The minimum value for each answer result is 1, indicating "no", and the maximum value is 4, indicating "very much". Higher scores on the functional scales/items indicate better functional status. Higher scores on the symptom scales/items indicate more severe symptoms. Higher scores on the global health status/QoL scale indicate better global health status/QoL.
Device performance evaluation | On the day of the ablation procedure
  Device performance of the investigational medical devices Navigational Bronchoscopy System and Bronchoscope and Accessories is evaluated by the treating investigator on the day of the ablation procedure.
  The highest score is 5, indicating excellent performance, while the lowest score is 1, signifying poor performance. Higher scores on the device performance evaluation indicate better device performance.

OTHER OUTCOMES:
Adverse events (AEs) / Serious Adverse Events (SAEs) | * Screening period/ Baseline (Day -30 to Day 0) * Treatment period / the day of ablation procedure (Day 0) * Day 1 post-treatment, within 24 hours after treatment * 1 month post-treatment * 3 months post-treatment
  Observe whether there are AEs or SAEs throughout the trial, count the number of cases and events and calculate the incidence (%).
Device-related AEs / device-related SAEs | * Treatment period / the day of ablation procedure (Day 0) * Day 1 post-treatment, within 24 hours after treatment * 1 month post-treatment * 3 months post-treatment
  Observe whether there are device-related AEs or SAEs throughout the trial, count the number of cases and events and calculate the incidence (%).
Complications | * Treatment period / the day of ablation procedure (Day 0) * Day 1 post-treatment, within 24 hours after treatment * 1 month post-treatment * 3 months post-treatment
  Observe whether there are complications during the clinical trial, count the number of cases and events and calculate the incidence (%).
  Complications include but not limited to: pneumothorax, pleural effusion, hemorrhage (intrapulmonary hemorrhage/hemothorax), pulmonary infection, cavity formation, and other rare complications (bronchopleural fistula, acute respiratory distress syndrome, non-target area frostbite, rib fracture, cold shock, thrombocytopenia, tumor needle tract implantation, nerve injury (brachial plexus, intercostal, phrenic, recurrent laryngeal nerves, etc.), pulmonary embolism, air embolism, cardiac tamponade, etc.) .

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Principal Investigator — Shanghai Chest Hospital; Calvin Ng, Principal Investigator — Chinese University of Hong Kong, Prince of Wales Hospital
Locations (2):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China
- Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No